CLINICAL TRIAL: NCT04662463
Title: Evaluation of Parturients With Anxiety
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting patients.
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Jie Zhou, Assistant Professor, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017P000696
Record Dates: First submitted 2018-07-31; First posted 2020-12-10 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBM-I assignment (Experimental): Patients will receive CBM-I assignments
  Interventions: Behavioral: Cognitive Bias Modification for Interpretation (CBM-I)
- Placebo assignment (Placebo Comparator): Patients will receive placebo assignments
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Cognitive Bias Modification for Interpretation (CBM-I) — Patients will receive CBM-I training by reading and imaging themselves in a series of emotionally ambiguous scenarios. Each scenario ends with an incomplete final word. Patients need to complete the final word to resolve the scenario in a positive direction.
  Arms: CBM-I assignment
Behavioral: Placebo — Patients will receive placebo task which uses neutral rather than emotional material.
  Arms: Placebo assignment

SUMMARY:
The primary objective of this study is to examine the effects of cognitive bias modification for interpretation (CBM-I) on prenatal anxiety in parturients. Half of the participants will receive CBM-I assignments, while the other half will receive placebo assignments.

DETAILED DESCRIPTION:
Maternal prenatal anxiety has been shown to have implications on neonatal behavior and early childhood behavioral and emotional wellbeing. Recent studies found that adults using computer-assisted feedback-learning paradigms, referred to as Cognitive Bias Modification for Interpretation (CBM-I), experienced significant reductions in levels of social anxiety, trait anxiety, and depression. Our goal is to identify patients with prenatal anxiety and evaluate the effects of CBM-I on symptoms of prenatal anxiety and patient satisfaction with the labor and delivery experience.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* Women before 36-week gestation
* At least high school level education

Exclusion Criteria:

* They refuse
* Have impaired decision-making capacity
* Are blind or extremely visually impaired (excluding use of glasses)
* Cannot understand or read English
* Diagnosed with psychiatric disorder other than anxiety

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Parturients only
Enrollment: 0 (Actual)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Effects of Internet-Based Cognitive Bias Modification (CBM-I) on prenatal anxiety | 4 weeks (starting from 36-week gestation)
  Change in State-Trait Anxiety Inventory (STAI) scores before and after the CBM-I assignment.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Zhou, MD, MS, MBA, Principal Investigator — Harvard Medical School (HMS and HSDM)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lester KJ, Field AP, Muris P. Experimental modification of interpretation bias about animal fear in young children: effects on cognition, avoidance behavior, anxiety vulnerability, and physiological responding. J Clin Child Adolesc Psychol. 2011;40(6):864-77. doi: 10.1080/15374416.2011.618449. PMID 22023278
- [Result] Bowler JO, Mackintosh B, Dunn BD, Mathews A, Dalgleish T, Hoppitt L. A comparison of cognitive bias modification for interpretation and computerized cognitive behavior therapy: effects on anxiety, depression, attentional control, and interpretive bias. J Consult Clin Psychol. 2012 Dec;80(6):1021-33. doi: 10.1037/a0029932. Epub 2012 Sep 10. PMID 22963595
- [Result] O'Connor TG, Ben-Shlomo Y, Heron J, Golding J, Adams D, Glover V. Prenatal anxiety predicts individual differences in cortisol in pre-adolescent children. Biol Psychiatry. 2005 Aug 1;58(3):211-7. doi: 10.1016/j.biopsych.2005.03.032. PMID 16084841